CLINICAL TRIAL: NCT03041818
Title: Development of Horse-Riding Program Model for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Konkuk University (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Bo Young Hong, Assistant professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 316086-2
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Cerebral Palsy; Motor Activity
Keywords: cerebral palsy; horseback riding
MeSH Terms: conditions — Cerebral Palsy; Motor Activity | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hippotherapy (Experimental): 16 sessions of horseback riding therapy
  Interventions: Behavioral: Horseback riding therapy

INTERVENTIONS:
Behavioral: Horseback riding therapy — Apply 30 minutes/session, twice a week for 8 weeks of horseback riding therapy (provided with 1 horse rider, 2 side walkers)
  Other Names: hippotherapy

SUMMARY:
The purpose of this study is to develop healing riding algorithm applicable in rural riding centers and to apply this to children with cerebral palsy.

DETAILED DESCRIPTION:
Horseback riding activities in Korea's riding centers have mostly centered on physical rehabilitation for children with special needs, including those with cerebral palsy, mental disabilities, and autism, with the program conducted by certified equine-assisted therapy instructors. However, there is no definite way to assess the ability of children for horseback riding and no standard riding program. Therefore, developing a assessment and program algorithm for healing horseback riding is expected to contribute to providing more activities for children with special needs and also for general people.

Children older than 4 years old or adolescent with cerebral palsy who voluntarily want to enroll this study would be enrolled.

Participants have 2 times of 30-minute horse riding program for 8 weeks, total 16 times of riding program in a local horse riding center.

Sample size assessment: Calculating for 20% of drop out, 16 patients were calculated to apply the assessment and applicable program.

Drop out: missing more than 2 lessons of horse-riding

Plan for missing data: not included

Statistical analysis plan: paired t-test for the outcome measures

ELIGIBILITY:
Inclusion Criteria:

* Children or adolescent with cerebral palsy
* GMFCS level I, II, III
* Body weight less than 80 kg

Exclusion Criteria:

* Medical condition who are not suitable for hippotherapy: severe osteoporosis, mental illness, not controlled seizure disorder etc.
* Social condition who are not suitable for hippotherapy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change of gross motor function (assessment of GMFM-88) | Before the program starts (up to 2 weeks), After the program ends (up to 2 weeks)
  Assessment of GMFM-88 before and after the 16 sessions of horse riding program
Change of Berg balance (assessment of pediatric berg balance scale) | Before the program starts (up to 2 weeks), After the program ends (up to 2 weeks)
  Assessment of pediatric berg balance scale before and after the 16 sessions of horse riding

SECONDARY OUTCOMES:
Actigraph (to monitor activity) | During the horse riding therapy/
  wear an Actigraph to monitor activity of children
Child Health Questionnaire (CHQ) | Before the program starts (up to 2 weeks), After the program ends (up to 2 weeks)
  Caregivers answer the sheets
Postural Assessment Scale for Hippotherapy (PASH) | From starting the therapy, every 2 weeks re-evaluated through study completion, in total 4 times
  Developed tool for assessment of ability for hippotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Bo Young Hong, MD, Principal Investigator — St.Vincent's hospital, The Catholic University of Korea
Locations (1):
- St. Vincent's hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: Yes
1 professor in Samsung Medical Center
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: When analysis is done after completion of the study
Access Criteria: Primary investigator of the study